CLINICAL TRIAL: NCT01899430
Title: Short-term Liraglutide Treatment in Obese Women With Polycystic Ovary Syndrome
Brief Title: Polycystic Ovary Syndrome and Liraglutide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, professor, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120047
Record Dates: First submitted 2013-07-07; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: PCOS; Obesity
Keywords: PCOS; obesity; GLP-1 receptor agonist; liraglutide; metformin
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Solutions; Injections; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Active Comparator): In the MET group metformin was initiated at a dose of 500 mg once per day and increased by 500 mg every 3 days up to 1000 mg BID per os.
  Interventions: Drug: metformin
- liraglutide (Experimental): In the LIRA group liraglutide was initiated at a dose of 0.6 mg injected sc once per day and increased to 1.2 mg/day after 1 week.
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide
  Other Names: Victoza 6 mg/ml solution for injection in pre-filled pen
  Arms: liraglutide
Drug: metformin
  Other Names: Glucophage tablets
  Arms: metformin

SUMMARY:
The purpose of this study was to determine whether liraglutide is more effective than metformin in the treatment of obese women with newly diagnosed polycystic ovary syndrome (PCOS). We anticipated greater changes in body weight in patients treated with liraglutide than in those treated with metformin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (NICHD criteria)
* BMI of 30 kg/m² or higher

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* history of carcinoma
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of MEN 2
* significant cardiovascular, kidney or hepatic disease
* the use of medications known or suspected to affect reproductive or metabolic functions
* the use of statins, within 90 days prior to study entry

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in body weight. | Patient's body weight was mesured at the base point and every four weeks during 12 weeks of clinical trial.

SECONDARY OUTCOMES:
The secondary outcome was change in body mass index (BMI) | Patient's body weight were measured at the base point and every four weeks during the 12 weeks of clinical trial. Patient's height was measured at the basepoint.
  Patient's BMI was defined as the patient's body mass in kilograms divided by the square of their height in meters.
The secondary outcome was change in waist circumference. | Patient's waist circumference was measured at the basepoint and every four weeks during 12 weeks of clinical trial.
  Patient's waist circumference was measured in centimeters.

OTHER OUTCOMES:
The other outcomes was changes changes in fasting concentrations of glucose. | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting glucose was measured in mmol/L.
Other outcome was change in fasting concentration of insulin. | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Fasting concentrations of insulin was measured in mU/L.
Other outcome was change in blood concentrations of LH (luteinizing hormone). | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Comncetration of LH was measured in U/L.
Other outcome was change in blood concentrations of FSH (follicle-stimulating hormone). | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of FSH was measured in U/L.
Other outcome was change in blood concentration of testosterone. | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentration was measured in nmol/L.
Otehr outcome was change in blood concentration in androstenedione. | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of androstenedione was measured in nmol/L.
Other outcome was change in blood concentrations of SHBG (sex hormone-binding globulin). | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of SHBG was measured in nmol/L.
Other outcome was change in blood concentration of DHEAS (dehydroepiandrosterone sulfate) | Patient's fasting blood was drawn at the basepoint and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of DHEAS was measured in micromol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia